CLINICAL TRIAL: NCT00273286
Title: Family Management of Childhood Diabetes Study
Brief Title: Family Management of Type 1 Diabetes in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Tonja Nansel, Eunice Kennedy Shriver National Institute of Child Health and Human Development
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMOD
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Insulin-Dependent; Diabetes Mellitus, Juvenile-Onset; IDDM; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- family diabetes management intervention (Experimental): A trained health advisor will be responsible for interactions with parents and patients prior to each diabetes clinic visit (Preparation Phase), at the time of the diabetes clinic visit (Consolidation Phase) and by phone, e-mail, etc. after the clinic visit (Follow-up Phase). Using educational modules developed for the study, families will be engaged in problem identification and solving activities to improve shared parent-youth responsibility for diabetes management and foster increased adolescent's independent management capabilities.
  Interventions: Behavioral: family diabetes management intervention

INTERVENTIONS:
Behavioral: family diabetes management intervention — a clinic-integrated, low intensity, multi-component behavioral intervention

SUMMARY:
This is a multi-center, randomized controlled trial to test whether a clinic-integrated, low intensity, multi-component behavioral intervention is effective in preventing the deterioration in glycemic control, treatment adherence, and quality of life that commonly occur during late childhood and early adolescence in youth with type 1 diabetes. The study will also examine mechanisms and processes that influence the effectiveness of family management of diabetes during this developmental period.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of a practical, low-cost, low-intensity behavioral intervention that can be integrated directly into diabetes clinic routines. The goal of the intervention is to prevent the deterioration in glycemic control, treatment adherence, and quality of life that often occur during the transition to adolescence in families of youth with type 1 diabetes. Four-hundred and eighty families (120 from each of the four sites) will be randomly assigned by the coordinating center to intervention or standard care conditions. Standard care will be the multidisciplinary management of type 1 diabetes as currently practiced at the clinical sites. Randomization will be stratified by main versus recent-onset subgroup, age, and for the main subgroup, baseline glycosylated hemoglobin level. Families will remain in their respective experimental conditions for 24 months. A trained health advisor will be responsible for interactions with parents and patients prior to each diabetes clinic visit (preparation phase), at the time of the diabetes clinic visit (consolidation phase) and by phone, e-mail, etc. after the clinic visit (follow-up phase). Using educational modules developed for the study, families will be engaged in problem identification and solving activities to foster improved disease management capabilities and improved parent-youth communication around and sharing of responsibility for diabetes management. Families will be assessed at home three times and in the clinic four times over the course of the study. Measures include parent, child, and family characteristics that may affect intervention effectiveness, targeted mediators, family interaction, management practices, and glycosylated hemoglobin (HbA1c). Primary outcomes are diabetes management adherence and metabolic control; secondary outcomes are quality of life, health status, and psychosocial status.

ELIGIBILITY:
Child Inclusion Criteria:

* Age 9.0 to <14.5.
* Type 1 diabetes diagnosis (diagnosed by ADA criteria) for a minimum of 1 year for the main subgroup or 3 months for the recent onset subgroup.
* Insulin dose greater than or equal to 0.5 u/kg/day for the main subgroup or 0.2 u/kg/day for the recent onset subgroup; with 2 or more daily injections or use of insulin pump.
* Most recent A1c is >6.0% and <13.0%; <12.0% for those diagnosed for less than 1 year.
* Willing to provide informed assent.

Parent/Family Environment Inclusion Criteria

* Child lives in geographically stable home, no multiple foster homes, boarding school, or institutions expected in next 2 years.
* The same 1 or 2 adult caregivers have accompanied the child to every diabetes clinic visit in the past year, and at least 1 caregiver agrees to participate in all aspects of the protocol (single-parent families, blended families, and separated parents will be eligible).
* Home has telephone access.
* Child had at least 2 clinic visits within last 12 months.
* Parent and child willing to come to clinic every 3 months for duration (2 years) of study.
* If a family has more than one eligible child, all qualifying children who provide consent/assent will participate in assessment and intervention or control activities; however, only the oldest qualifying child will be included in statistical analyses.

Child Exclusion Criteria:

* Presence of a major chronic diseases (except well-controlled thyroid, asthma, celiac).
* Presence of a major visual/auditory impairments.
* Child is in a self-contained special education class throughout the school day.
* Record of inpatient hospitalization for mental disorder in past six months including substance abuse rehabilitation, eating disorder units or day treatment programs. Current diagnosis of eating disorder. History of anti-psychotic medications for the past 6 months.
* Diagnosis of mental retardation.
* Unable to read and write English at 2nd grade level.
* Children who are currently enrolled in any intervention study are not eligible for enrollment. Those who have been in an intervention arm of a trial of a behavioral, psychological or psychoeducational intervention and concluded their study follow-up within the past 12 months are also ineligible to participate. However, children who were in a standard care control group in an intervention study are eligible once they have completed all scheduled study follow-ups. Children cannot enroll in another intervention study during the course of this study. Enrollment of children who are currently participating in another observational study will be at the discretion of the site principal investigator.

Parent/Family Environment Exclusion Criteria

* Family has plans to re-locate out of area within the next 2 years of the study.
* Participating caretaker is currently undergoing treatment for substance abuse.
* Participating caretaker has been hospitalized in past 6 months for mental disorder.
* Participating caretaker has history of psychosis.
* Families who are currently enrolled in any intervention study are not eligible for enrollment. Those who have been in an intervention arm of a trial of a behavioral, psychological or psychoeducational intervention and concluded their study follow-up within the past 12 months are also ineligible to participate. However, families who were in a standard care control group in an intervention study are eligible once they have completed all scheduled study follow-ups. Families cannot enroll in another intervention study during the course of this study. Enrollment of families who are currently participating in another observational study will be at the discretion of the site principal investigator.

The family must reside within 90 miles (one-way) of the clinic (main or satellite), or agree to meet at a mutually agreed upon closer location for conduct of the home assessment.

Ages: 108 Months to 174 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 422 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
glycemic control | 1/2006-3/2009
  HbA1c
treatment adherence | 1/2006-3/2009
  Diabetes Self Management Profile

SECONDARY OUTCOMES:
quality of life | 1/2006-3/2009
  PedsQL Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Simons-Morton, PhD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (4):
- United States (4):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Temmen CD, Lu R, Gee BT, Chen Z, Nansel TR. Latent classifications of parental involvement in diabetes management for youth with type 1 diabetes: A randomized clinical trial. Pediatr Diabetes. 2022 Nov;23(7):1133-1142. doi: 10.1111/pedi.13397. Epub 2022 Aug 19. PMID 36250647
- [Derived] Nansel TR, Thomas DM, Liu A. Efficacy of a Behavioral Intervention for Pediatric Type 1 Diabetes Across Income. Am J Prev Med. 2015 Dec;49(6):930-4. doi: 10.1016/j.amepre.2015.05.006. Epub 2015 Jul 29. PMID 26231856
- [Derived] Nansel TR, Lipsky LM, Iannotti RJ. Cross-sectional and longitudinal relationships of body mass index with glycemic control in children and adolescents with type 1 diabetes mellitus. Diabetes Res Clin Pract. 2013 Apr;100(1):126-32. doi: 10.1016/j.diabres.2012.12.025. Epub 2013 Jan 20. PMID 23339757
- [Derived] Nansel TR, Iannotti RJ, Liu A. Clinic-integrated behavioral intervention for families of youth with type 1 diabetes: randomized clinical trial. Pediatrics. 2012 Apr;129(4):e866-73. doi: 10.1542/peds.2011-2858. Epub 2012 Mar 5. PMID 22392172